CLINICAL TRIAL: NCT05552521
Title: Early Diastolic Dysfunction in Patients With Septic Shock and Its Association With the Presence of Cardiomyopathy Genetic Variants
Brief Title: Diastolic Dysfunction in Septic Shock and Cardiomyopathy Genetic Variants
Acronym: SepticHeartG
Status: Completed | Type: Observational
Sponsor: Hospital Garcia de Orta (Other)
Collaborators: Instituto de Medicina Molecular João Lobo Antunes (Other)
Responsible Party: Principal Investigator, Filipe André Gonzalez, Senior consultant of Internal Medicine and Intensive Medicine, PhD student, Hospital Garcia de Orta
Other Study IDs: TI 01/2022
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Diastolic Dysfunction; Septic Shock; Cardiomyopathies
MeSH Terms: conditions — Shock, Septic; Cardiomyopathies | interventions — Echocardiography; Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For genetic analysis, blood will be withdrawn from patients at ICU admission and sent to a certified laboratory for whole-exome sequencing in collaboration with the Institute of Molecular Medicine (IMM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography in 4 timepoints: 1st 24h + 7th-10th day; 28th-30th day; 6 months Whole exome sequencing at admission
  Other Names: Genetic analysis

SUMMARY:
Sepsis is a life-threatening infection with increasing incidence, and its spectrum of disease can involve cardiac dysfunction, which further adds to mortality. Although cardiac involvement in sepsis has been classically attributed to systolic dysfunction, diastolic dysfunction is increasingly diagnosed due to new echocardiographic techniques and the conceptual evolution of diastolic dysfunction. Combining systolic and diastolic dysfunction assessment could lead to a better diagnosis of septic cardiac dysfunction. Furthermore, earlier forms of septic cardiac dysfunction could be more promptly recognized by measuring novel and less used parameters of diastolic dysfunction. We hypothesize that left atrium (LA) strain and isovolumetric relaxation time (IVRT) derived intervals could be new and earlier predictors of diastolic dysfunction in septic patients with a potential impact on clinical presentation and prognosis and that rare genetic variation associated with inherited cardiomyopathies could underline the risk and severity of sepsis-related myocardial dysfunction with potential impact on diagnosis and prognosis.

DETAILED DESCRIPTION:
Primary outcome:

Presence of diastolic dysfunction at baseline or during evolution in patients presenting with septic shock and its impact on prognosis.

Secondary outcomes:

Development of heart failure symptoms and presence of myocardial dysfunction (either systolic or diastolic) at 30th day, 30-day mortality, mechanical ventilation duration, ICU length of stay, and hospital stay, and need for therapeutic change.

Mid-term prognosis will be assessed at six months follow-up for evaluation of the clinical functional class, LV systolic and diastolic function, and biomarkers.

METHODS AND TASK DESCRIPTION A prospective multicenter observational study in the 24-bed polyvalent ICU of Hospital Garcia de Orta, Almada, Portugal. Expected sample size of 140 patients, to have a confidence level of 95%, with a precision within ± 5% (population of septic patients in the ICU/yearly).

Population :

* Inclusion: All patients admitted in the ICU i. ≥ 18 years old; ii. with septic shock by the sepsis 3.0 criteria: Sepsis and (despite adequate volume resuscitation) both of: persistent hypotension requiring vasopressors to maintain MAP greater than or equal to 65 mm Hg, and lactate greater than or equal to 2 mmol/L.
* Exclusion: pregnancy, congenital heart disease, artificial valve prosthesis, severe aortic or mitral pathology, atrial fibrillation, and inadequate image quality.

Study design summary A comprehensive echocardiogram is performed by an intensive care and echocardiography specialist at five-time points: the earliest opportunity following admission (< 24h); from 3rd to 5th day; from 7th to 10th day; 28th to 30th day or at ICU discharge, if before; and at 6-month (either in hospital or ambulatory) and at 28th day. Also, invasive arterial pressure and central venous pressure, and cardiac biomarkers (highly sensitive troponin T and NT-proBNP) will be measured in all the timepoints, and inflammatory biomarkers (adrenomedullin, IL-1 and 6) will be measured at baseline, between day 7 and 10, and at 28th day or discharge and at 6 months.

Echocardiography All echocardiographic measures are obtained with simultaneous ECG display, and the three different sets of measures are obtained with the patient in the same position. All Doppler measurements are averaged from three measurements in sinus rhythm.

In addition to the qualitative examination of chambers and valves, the following measurements are obtained via the standard parasternal and apical views:

* Pulmonary Artery Systolic Pressure: If the patient has tricuspid regurgitation, measured by continuous Doppler in Parasternal short axis, Parasternal view of right ventricular inflow tract or Apical four Chamber view.
* Left Atrium Measurements: Size, (M-Mode, 2D) Volume, in Apical 4 Chamber view and Apical 2 Chamber view).
* Left and Right Ventricle 2D Color and Doppler: LV end-diastolic and end-systolic volumes (EDV and ESV) using biplane modified Simpson's rule, from which EF is calculated; RV end-diastolic area ratio Fractional Area Change (FAC) of RV and Tricuspid Annular Plane Systolic Excursion (TAPSE); LVOT diameter, LVOT VTI measured on pulsed-wave Doppler from which SV is calculated. Then CO and CI derived at inspiration and expiration.
* Mitral Flow Measurements: E maximal velocity, A maximal velocity. 4-Chamber apical view, Pulsed Doppler, Average of 3 measurements in SR. Isovolumetric relaxation time, isovolumetric contraction time, and ejection time are measured on pulsed-wave Doppler in apical five-chamber, and care is taken to display distinct aortic valve closure and mitral valve opening signals simultaneously, and then MPI is derived, normalized to heart rate.
* Tissue Doppler Measurements: RV S wave, Septal e' and Lateral e' on four-chamber apical view. Average of 3 measurements in SR. The myocardial isovolumic relaxation time (IVRT') is measured from the end of systolic myocardial velocity during ejection (Sa) to onset of the early diastolic myocardial velocity (e') at the left lateral and septal mitral annulus, and the average is used; the time difference IVRT-IVRT' is further calculated to obtain the [IVRT-IVRT'] parameter. Myocardial Performance Index (MPI) is also calculated.
* Left Ventricular and Left Atrial strain: Images are analyzed offline using dedicated software. Global Longitudinal Strain is calculated as the average speckle tracking strain from each of the 18 LV segments from the 2, 4, and 3-chamber views. Peak strain value is derived from the maximal inflection point on the composite LA strain curve and grade based on recently published cutoffs. Calculations of LA functionality to assess conduit, reservoir, and booster function is performed using definitions from previous studies.

Tissue Doppler measurements are taken from the modal velocity, from septal and lateral mitral annulus.

Systolic dysfunction is defined as those with a calculated EF < 50%. Diastolic dysfunction is classified according to 2016 ASE/EACVI guidelines with a focused analysis on the simplified criteria as E/e' >15 and e' < 0.08 m/s.

Repeated measures for different echocardiographic parameters are taken by the same physician and by two different physicians to assess inter-and intra-observer variability.

Genetic analysis For genetic analysis, blood will be withdrawn from patients at ICU admission and sent to a certified laboratory for whole-exome sequencing, in collaboration with the Institute of Molecular Medicine (IMM).

Hemodynamic monitoring Continuous hemodynamic monitoring will be achieved by a bioimpedance device - Starling Baxter - in the first 72 hours, for registration of the following variables: indexed stroke volume, stroke volume variation, cardiac output, cardiac index, heart rate, dX/dt, ventricular ejection time, total fluid content (and the dynamic variation), total peripheral resistance index and cardiac power index.

Clinical data and biochemical biomarkers All demographic, clinical, hemodynamic, respiratory data, fluid balance, vasopressors, and lab results - including highly sensitive troponin T, NT-proBNP, adrenomedullin, IL-1, and 6 - are prospectively collected, as well as SOFA, SAPS-II, APACHE-II scores, and mortality until 30 days and 6-month of follow-up.

Statistics Continuous variables are expressed as mean ± standard deviation or median and interquartile range and compared between any two groups using t-test or the Mann-Whitney U test, as appropriate. The normality of distribution is evaluated by visual inspection of histograms and by the Kolmogorov Smirnov test. Categorical variables are expressed as proportions and compared with the Mantel- Haenszel Chi-square test or Fisher exact test.

A mathematical model (curve and surface fitting, and time series regression) will be created so that the LA strain rate and IVRT variables could be predictors of early diastolic dysfunction. Associations between rare genetic variants and the development of early and late cardiac dysfunction are tested.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the ICU i. ≥ 18 years old; ii. with septic shock by the sepsis 3.0 criteria (13): Sepsis and (despite adequate volume resuscitation) both of: persistent hypotension requiring vasopressors to maintain MAP greater than or equal to 65 mm Hg, and lactate greater than or equal to 2 mmol/L.

Exclusion Criteria:

* pregnancy, congenital heart disease, artificial valve prosthesis, severe aortic or mitral pathology, atrial fibrillation, and inadequate image quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective multicenter observational study in the 30-bed polyvalent ICU of Hospital Garcia de Orta, Almada, Portugal. Expected sample size of 140 patients, to have a confidence level of 95%, with a precision within ± 5% (population of septic patients in the ICU/yearly).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Diastolic dysfunction | through study completion until 6 months
  Left atrium strain in % and IVRTs intervals in msec
Hereditary Cardiomyopathy genetic variants | through study completion until 6 months
  Search for cardiomyopathies genetic variantes that could explain a myocardial susceptibility to develop injury in septic shock

SECONDARY OUTCOMES:
Heart failure | through study completion until 6 months
  heart failure symptoms according to NYHA clarification at 30 days and 6 months
Mortality | through study completion until 6 months
  Mortality at 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Filipe A Gonzalez, MD, PhD st., Principal Investigator — Hospital Garcia de Orta
Locations (1):
- Hospital Garcia de Orta, Lisbon, Almada, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Walley KR. Sepsis-induced myocardial dysfunction. Curr Opin Crit Care. 2018 Aug;24(4):292-299. doi: 10.1097/MCC.0000000000000507. PMID 29846206
- [Background] Landesberg G, Gilon D, Meroz Y, Georgieva M, Levin PD, Goodman S, Avidan A, Beeri R, Weissman C, Jaffe AS, Sprung CL. Diastolic dysfunction and mortality in severe sepsis and septic shock. Eur Heart J. 2012 Apr;33(7):895-903. doi: 10.1093/eurheartj/ehr351. Epub 2011 Sep 11. PMID 21911341
- [Background] Rapezzi C, Arbustini E, Caforio AL, Charron P, Gimeno-Blanes J, Helio T, Linhart A, Mogensen J, Pinto Y, Ristic A, Seggewiss H, Sinagra G, Tavazzi L, Elliott PM. Diagnostic work-up in cardiomyopathies: bridging the gap between clinical phenotypes and final diagnosis. A position statement from the ESC Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 May;34(19):1448-58. doi: 10.1093/eurheartj/ehs397. Epub 2012 Dec 4. PMID 23211230
- [Derived] Gonzalez FA, Bacariza J, Varudo AR, Leote J, Mateus RM, Martins CM, Ribeiro MI, Sanfilippo F, Lopes LR, Almeida AG. Sepsis-induced myocardial dysfunction diagnosed with strain versus non-strain echocardiography parameters: incidence, evolution and association with prognosis. Ann Intensive Care. 2025 Sep 25;15(1):141. doi: 10.1186/s13613-025-01561-w. PMID 40999250